CLINICAL TRIAL: NCT00632905
Title: A Prospective Study to Evaluate the Incidence of Skeletal Related Events In Prostate Cancer Patients Undergoing Androgen Deprivation Therapy (ADT).
Brief Title: Bone Health Observational Study
Acronym: BHOS
Status: Completed | Type: Observational
Sponsor: CMX Research (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: AZ-CMX-03
Record Dates: First submitted 2008-02-20; First posted 2008-03-11 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostatic adenoma; Prostatic neoplasm
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Normal - BMD with T-score at or above -1.0
- 2: Osteopenic - BMD with T-score between -1.1 and -2.4
- 3: Osteoporotic - BMD with T-score at or below -2.5

SUMMARY:
Prostate Cancer patients treated with LHRH agonists (e.g., goserelin) lose Bone Mineral Density (BMD). Using a prospective, observational study design, we propose that monitoring how physicians manage Cancer Treatment Induced Bone Loss(CTIBL) in their patients. The gold standard for evaluating BMD is dual energy x-ray absorptiometry (DEXA). The proposed study will provide some of the first prospective data on the rates of Skeletal Related Events (SREs) in prostate cancer patients undergoing ADT and help develop official guidelines on the use of DEXA screening for prostate cancer patients.

DETAILED DESCRIPTION:
A consequence of ADT is the gradual bone loss, so-called cancer treatment induced bone loss (CTIBL). The current standard of care is the addition of Vitamin D and Calcium upon the initiation of ADT. Moreover, bisphosphonates are now being considered to treat and prevent CTIBL. However, bisphosphonates are costly, thus there is a desire to identify or target a specific subset of patients who would most benefit from the treatment.

By obtaining baseline BMD and monitoring for Skeletal Related Events (SREs), we hope to identify that specific sub-set of patients who would most benefit from the treatment. Using a prospective, observational study design, we propose monitoring how physicians manage CTIBL in their patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to provide written Informed Consent.
* Patients for whom Androgen Deprivation Therapy (ADT) with Zoladex® is indicated for at least 1 year.
* Patients started on Zoladex® within the last 4 months.

Exclusion Criteria:

* Patient had surgery or significant traumatic injury occurring within 1 month prior to consent.
* Known hypersensitivity to Goserelin Acetate or any of the components found in Zoladex®.
* Any concurrent condition that would make it undesirable, in the physician's opinion, for the subject to participate in the study or would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2007-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density of the lumbar spine | 12 months

SECONDARY OUTCOMES:
Overall Safety | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Casey, M.D., Principal Investigator — CMX Research
Locations (40):
- Canada (40):
  - Dr. John A. Warner, Burnaby, British Columbia
  - Southern Interior Medical Research Corporation, Kelowna, British Columbia
  - Nanaimo Urology Associates, Nanaimo, British Columbia
  - Central Island Research Centre, Port Alberni, British Columbia
  - Andreou Research, Surrey, British Columbia
  - Bruce W. Palmer Urology Inc., Kentville, Nova Scotia
  - Dr. Jonathan L. Giddens, Brampton, Ontario
  - Brantford Urology Research Medical Arts Bldg., Brantford, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Dr. Richard Sowery, Burlington, Ontario
  - Northern Urology Centre, Greater Sudbury, Ontario
  - Guelph Urology Associates, Guelph, Ontario
  - Dr. Alvaro Morales, Kingston, Ontario
  - GU Trials Markham, Markham, Ontario
  - Mor Urology Inc, Newmarket, Ontario
  - Medical & Dental Bldg, North Bay, Ontario
  - Stanley Flax Medicine Professional Corporation, North York, Ontario
  - York-Finch Med Centre, North York, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - Orillia Urology Associates, Orillia, Ontario
  - Urotec, Oshawa, Ontario
  - Mahoney Medicine Professional Corporation, Ottawa, Ontario
  - 2150935 Ontario Inc, Owen Sound, Ontario
  - Kawartha Urology Associates, Peterborough, Ontario
  - The Medical Centre, Peterborough, Ontario
  - Dr. Allan Abramovitch, Scarborough Village, Ontario
  - Dr. Peter Roney, Smiths Falls, Ontario
  - West Arthur Place, Thunder Bay, Ontario
  - Dr. Edward Woods, Toronto, Ontario
  - The Male Health Centre, Toronto, Ontario
  - Dr. Roger Buckley, Willowdale, Ontario
  - ABHM Associates, Windsor, Ontario
  - Dr. Louis-Rene Barrette, Chicoutimi, Quebec
  - Recherches Cliniques Theradev, Granby, Quebec
  - Polyclinique Med Concorde, Laval, Quebec
  - Ultra-Med Inc., Point Claire, Quebec
  - Clinique d'Urologie du Saguenay, Saguenay, Quebec
  - Centre de Récherche en Urologie de Lanaudiére, Saint Charles-Baromee, Quebec
  - Westmount Med Bldg, Westmount, Quebec
  - Medical Arts Bldg, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided